CLINICAL TRIAL: NCT00908999
Title: FMRI of Anosognosia in Amnestic MCI and AD: Focus on Cortical Midline Structures
Brief Title: Functional Magnetic Resonance Imaging (fMRI) of Anosognosia in Amnestic Mild Cognitive Impairment (MCI) and Alzheimer's Disease (AD)
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: HSC-2008-0090
Record Dates: First submitted 2009-05-22; First posted 2009-05-27 (Estimated); Last update posted 2011-09-29 (Estimated); Status verified 2011-09

CONDITIONS: Anosognosia; Alzheimer's Disease; Mild Cognitive Impairment
Keywords: anosognosia fMRI amnestic MCI Alzheimer; anosognosia in AD and MCI
MeSH Terms: conditions — Agnosia; Alzheimer Disease; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (3):
- Controls: The control group have to be medically and cognitively healthy(MMSE ≥ 28; Hopkins Verbal Memory Test-Revised raw score within 1.5 SD of normative values for age and gender). These individuals are recruited from the community and all attempts will be made to match them on age and education to individuals recruited for groups of AD and aMCI.
- amnestic Mild Cognitive Impairment: Participants who have expressed interest to take part in the study. A consensus from the study clinicians regarding the diagnosis will be required before a subject is enrolled. The criteria for MCI include 1) observation of memory decline by informant, 2) Mini Mental Status Exam (MMSE) score between 24 and 30, 3) objective memory impairment on neuropsychological tests, 3) intact functional abilities, and 4) no diagnosis of dementia.
- Alzheimer's disease: Patients with probable Alzheimer's disease according with the NINDS-ADRDA and DSM-IV diagnostic criteria. An additional criterion is a MMSE score between 16 and 27. All AD patients must have capacity to provide informed consent as judged by the referring physician.

SUMMARY:
This is a three year fMRI study conducted at the University of Wisconsin (UW) Hospital and the William. S. Middleton VA Hospital. This study is guided by the hypothesis that reduced fMRI activity and connectivity cortical midline structures (i.e., medial frontal and ventral posterior cingulate cortex) are physiologic abnormalities that relate strongly to the compromised insight into cognitive deficits, or anosognosia, shown by a subset of individuals with amnestic MCI (aMCI) and AD. Further, the investigators hypothesize that these regional changes in fMRI activity are predictive of faster progression from aMCI to AD.

ELIGIBILITY:
Inclusion Criteria:

* Amnestic MCI:

  1. Observation of memory decline by informant.
  2. Mini Mental Status Exam (MMSE) score between 24 and 30.
  3. Objective memory impairment on neuropsychological tests.
  4. Intact functional abilities, and 4) no diagnosis of dementia.
* AD:

  1. A diagnosis of probable AD according with the NINDS-ADRDA and DSM-IV diagnostic criteria.
  2. MMSE score between 16 and 27. All AD patients will have capacity to provide informed consent as judged by the referring physician.

Exclusion Criteria:

* MRI incompatibility; history of neurologic disease (including prior loss of consciousness of more than 10 minutes); prior neurosurgery; or chronic medical diseases (such as poorly controlled diabetes, renal disease, or poorly controlled hypertension).
* Excluded medications include neuroleptics, short or long acting nitrates, and Warfarin.
* Other exclusions include: less than 10 yrs of education; Hachinski scale of 4 or more; first language other than English; poor visual or auditory acuity; pregnancy.

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: MCI and AD patients are referred from memory clinics at the UW hospital, William S. Middleton Memorial Veterans Hospital (Madison, WI) and the statewide clinics offered through the Wisconsin Alzheimer's Institute (WAI).
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2008-04; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- William S Middleton VA Hospital GRECC, Madison, Wisconsin, United States